CLINICAL TRIAL: NCT04033705
Title: To Explore the Association Between Preoperative Indicators of Glycaemic Control and Perioperative Glycaemia Associated Risk in Patients With Type 2 Diabetes Undergoing Elective Orthopaedic Surgery Using Continuous Glucose Monitoring
Brief Title: DRIVE - Perioperative Period
Acronym: DRIVE-Periop
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/23
Record Dates: First submitted 2019-07-01; First posted 2019-07-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Surgical Procedure, Unspecified
Keywords: Perioperative; Continuous glucose monitoring; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Freestyle Libre Pro glucose sensor — Participants will wear a Freestyle Libre Pro glucose sensor for approximately 2 weeks prior to elective surgery and then for 2 weeks following surgery.

SUMMARY:
This study will investigate if the HbA1c result before surgery which assesses glucose control over the longer term, can accurately predict what happens to the glucose levels and glucose profile following surgery. This will be recorded using continuous glucose monitoring sensors which are worn by participants pre and post elective surgery.

DETAILED DESCRIPTION:
The research question addressed in this study is how preoperative markers of diabetes control correspond with the fluctuations in glucose levels which occur around surgery measured using continuous glucose monitoring (CGM). At present a HbA1c blood test prior to surgery is routinely used to infer the surgical risk associated with a person's glucose levels. HbA1c gives a measure of average blood glucose levels over the preceding 2-3 months and the joint British diabetes society guidelines recommend aiming for an HbA1c of 69mmol/mol or less before planned surgery.

However the HbA1c does not give a complete picture of a person's diabetes control and the evidence behind this threshold is incomplete. Furthermore due to the physiological stress of surgery and counterregulatory hormone release glucose levels can be more dynamic and unpredictable in this population. With CGM glucose levels are recorded multiple times an hour, revealing glucose variation and the amount of time the person's glucose levels spend above and below the ideal range which is understood to be associated with increased risks. This study aims to examine how such glucose patterns and 'at risk' time periods when glucose levels are outside of the target range correspond with different levels of HbA1c before surgery. This is an important area of study as diabetes is becoming increasingly prevalent in surgical patients and is associated with worse outcomes. Using new technologies to evaluate predictors of such harmful patterns in glucose levels is therefore vital.

Individuals who are eligible for this study are those with type 2 diabetes undergoing elective primary hip or knee replacement surgery. This is an observational study. Participants will wear a Freestyle Libre Pro glucose sensor for 2 weeks before and 2 weeks immediately post their surgery. The investigators will also collect information about participants recovery.

Duration of the study will be up to 8 weeks. The study will take place at Portsmouth Hospital NHS trust.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (on diet, oral, injectable and / or insulin therapy for diabetes)
* Be scheduled for primary elective hip or knee replacement surgery at Queen Alexandra Hospital
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Enrolled in another study that may affect glycaemic control over the 4-6 week period of active data collection with the sensor
* Taking oral steroids for longer than 2 weeks that incorporates the 4-6 week period of active data collection with the sensor
* Currently pregnant or planning pregnancy
* On dialysis
* Taking antipsychotic medication
* Non primary surgery (including emergency or revision surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who are undergoing elective primary total hip or knee replacement surgery at Queen Alexandra Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
The time spent within, above and below the target glucose range (4-10mmol/L) in the preoperative period | At week 2 following enrollment (this is pre surgery)
  The percentage of time spent within and outside of the target glucose range recorded by the glucose sensor
The time spent within, above and below the target glucose range (4-10mmol/L) in the post operative period | At week 4 following enrollment (this is post surgery)
  The percentage of time spent within and outside of the target glucose range recorded using the glucose sensor

SECONDARY OUTCOMES:
Length of hospital stay | This will be recorded at 2 weeks post surgery
  The number of days between hospital admission for elective surgery and the date of discharge
Post operative infections | This will be recorded at 6 weeks post surgery
  Investigators will record if the participant required antibiotics for infection from any source additional to those routinely prescribed as per hospital policy for the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kate Millar, MBChB, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No